CLINICAL TRIAL: NCT03093740
Title: Use of Direct-acting Antiviral Therapy to Prevent Spread of HCV Infection for Patients Receiving a HCV Positive Kidney Transplant as a HCV Negative Recipient
Brief Title: Direct-acting Antiviral Therapy to Prevent HCV Infection for HCV Positive Donor to HCV Negative Recipient Kidney Transplant
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrew IRB application, never approved and no subjects enrolled
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Raymond T. Chung, MD, Director, Hepatology, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000301
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Renal Failure Chronic; Hepatitis C
Keywords: hemodialysis; renal failure; kidney transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hepatitis C; Renal Insufficiency | interventions — elbasvir-grazoprevir drug combination; Sofosbuvir

STUDY DESIGN:
Intervention Model Description: Based on the genotype and viral resistance testing of the donor, that will be determined within the first week, we will initiate a genotype specific regimen for HCV treatment as available by prescription
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV treatment - no viral resistance (Experimental): Based on the genotype and negative viral resistance testing of the donor, (determined within the first week) we will initiate a genotype specific regimen of Zepatier
  Interventions: Drug: Zepatier
- HCV treatment - viral resistance (Experimental): Based on the genotype and positive viral resistance testing of the donor, (determined within the first week) we will initiate a genotype specific regimen of Zepatier plus Sofosbuvir
  Interventions: Drug: Zepatier plus Sofosbuvir

INTERVENTIONS:
Drug: Zepatier — Based on negative viral resistance testing of the donor treatment will be Zepatier
  Arms: HCV treatment - no viral resistance
Drug: Zepatier plus Sofosbuvir — Based on positive viral resistance testing of the donor treatment will be Zepatier with Sofosbuvir
  Arms: HCV treatment - viral resistance

SUMMARY:
Open label single center study for the donation of HCV positive kidneys to HCV negative recipients with interventional treatment to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
The study objective is to determine if the administration of direct acting antivirals for 12-16 weeks after kidney transplantation prevents the spread of HCV infection from donor kidney with known HCV infection (all genotypes) to an HCV negative recipient as evidenced by a negative HCV viral RNA at 12 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Donor meets MGH transplant center criteria and already listed for isolated kidney transplant
* No available living kidney donor
* Recipient has ≤ 730 days of accrued transplant waiting time
* Recipient chronic hemodialysis or peritoneal dialysis
* Recipient must agree to birth control.

  °.Weigh ≥ 50kg
* Serum ALT within normal limits
* Subject's Insurance company approves payment for DAA therapy post-kidney transplant

Exclusion Criteria:

* AB Blood type
* HCV genotype 1
* BMI > 35
* Any liver disease in recipient
* Pregnant or nursing (lactating) women
* Known allergy or intolerance to tacrolimus that would require administration of cyclosporine
* Albumin < 3g/dl or
* Platelet count < 75 x 103/mL
* Positive crossmatch or positive donor specific antibodies
* HCV RNA positive
* Hepatitis B surface antigen positive
* Patients with primary focal segmental glomerulosclerosis (FSGS)
* Any contra-indication to kidney transplantation per our center protocol

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Undetectable HCV RNA | 12 weeks post treatment
  Negative HCV viral load 12 weeks after last dose of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No current plans to share participant data